CLINICAL TRIAL: NCT04097886
Title: Investigating the Effects of Timed Exercise on Human Circadian Rhythms
Brief Title: Timed Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Pendergast (Other)
Responsible Party: Sponsor-Investigator, Julie Pendergast, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 45342
Record Dates: First submitted 2019-08-29; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Circadian Timing - Exercise
Keywords: circadian; phase shift; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Exercise Group (Experimental): Participants perform moderate exercise in the morning.
  Interventions: Other: Morning Exercise
- Evening Exercise Group (Experimental): Participants perform moderate exercise in the evening.
  Interventions: Other: Evening Exercise

INTERVENTIONS:
Other: Morning Exercise — moderate intensity exercise (70% VO2 max) each morning for 5 days
  Arms: Morning Exercise Group
Other: Evening Exercise — moderate intensity exercise (70% VO2 max) each evening for 5 days
  Arms: Evening Exercise Group

SUMMARY:
The purpose of this study was to investigate the effect of timed exercise on human circadian rhythms. Subjects were randomized to 5 days of morning or evening treadmill exercise. A measure of internal circadian timing, or phase, was measured at baseline and following the exercise intervention. Change in circadian phase was compared between the morning and evening group.

DETAILED DESCRIPTION:
This study investigated the effect of morning versus evening exercise on internal circadian timing, or phase. Young, sedentary subjects were recruited for this study. Baseline measures included anthropometric, body composition, cardiorespiratory fitness, chronotype, and circadian phase. Subjects were randomized to 5 consecutive days of morning or evening exercise. Thirty minutes of exercise was performed at the designated time and intensity was maintained at a heart rate corresponding with 70% peak VO2. The measure of circadian phase was salivary dim light melatonin onset, indicated by the time when saliva melatonin concentration exceeded 4pg/ml. Post-exercise circadian phase was measured the evening following the last day of exercise. Changes in circadian phase were compared between morning and evening groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-40.0
* sedentary; <=2 hrs structured exercise weekly
* medication free (other than birth control)

Exclusion Criteria:

* diagnosed conditions that would contraindicate safe participation in physical activity
* diagnosed psychiatric conditions
* night or rotating shift work 1-year prior to study
* travel across time zones within previous 4 weeks
* having children <2 years of age
* smoking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
Change in onset (time) of melatonin secretion | baseline and following completion of exercise intervention (approximately 5 days)
  Difference in onset (time at which salivary melatonin exceeds threshhold; 4pg/mL) from baseline to completion of exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Pendergast, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas JM, Kern PA, Bush HM, McQuerry KJ, Black WS, Clasey JL, Pendergast JS. Circadian rhythm phase shifts caused by timed exercise vary with chronotype. JCI Insight. 2020 Feb 13;5(3):e134270. doi: 10.1172/jci.insight.134270. PMID 31895695